CLINICAL TRIAL: NCT03423992
Title: A Pilot Study to Evaluate the Safety and Efficacy of Personalized Chimeric Antigen Receptor T Cell Immunotherapy for Patients With Recurrent Malignant Gliomas Based on the Expression of Tumor Specific/Associated Antigens
Brief Title: Personalized Chimeric Antigen Receptor T Cell Immunotherapy for Patients With Recurrent Malignant Gliomas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Mario Biotech Company (Unknown); Hebei Senlang BIotech Company (Unknown); Beijing HuiNengAn Biotech Company (Unknown)
Responsible Party: Principal Investigator, Qingtang Lin, Associate Professor, Department of Neurosurgery, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Xuanwu hospital
Record Dates: First submitted 2018-01-22; First posted 2018-02-06 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Glioma; Malignant Glioma of Brain; Recurrence Tumor
MeSH Terms: conditions — Glioma; Recurrence | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological: Chimeric antigen receptor T cells (Experimental)
  Interventions: Biological: chimeric antigen receptor T cells

INTERVENTIONS:
Biological: chimeric antigen receptor T cells — chimeric antigen receptor T cells expressing receptors specific for EGFRvIII, IL13Rα2, Her-2, CD133, EphA2, GD2, respectively

SUMMARY:
A pilot study to determine the safety and efficacy of chimeric antigen receptor T cell (autologous T cells transduced with a lentiviral vector expressing chimeric antigen receptor with or without anti-PDL1 antibody) personalized immunotherapy for patients with recurrent malignant gliomas based on the expression of tumor specific/associated antigens (EGFRVIII, IL13Rα2, Her-2, EphA2, CD133, GD2).

ELIGIBILITY:
Inclusion Criteria:

* Voluntary informed consent for entry of trial;
* Age greater than 18 years, and less than 70 years;
* Pathologically confirmed recurrent malignant gliomas;
* Tumor cells from resected tissue must be available for antigen testing (EGFRvIII, IL13Rα2, Her-2, CD133, EphA2, GD2) and at least one of the targets should be tested positively by immunohistochemistry study;
* If the patient is on dexamethasone, the anticipated dose must be 4 mg/day or less for at least 5 days prior to apheresis.
* Patients must have a Karnofsky performance status of greater than or equal to 70.
* Life expectancy greater than 3 months;
* Participants with adequate organ function as measured by:

  1. White blood count greater than or equal to 2500/mm^3; platelets greater than or equal to 100,000/mm^3, hemoglobin greater than or equal to 10.0 g/dL; without transfusion or growth factor support
  2. Aspartate transaminase (AST), Alanine transaminase (ALT), gamma glutamyl transpeptidase (GGT), lactic acid dehydrogenase (LDH), alkaline phosphatase within 2.5 x upper normal limit, and total bilirubin less than or equal to 2.0 mg/dL
  3. Serum creatinine less than or equal to 1.5 x upper limit of normal
  4. Coagulation tests prothrombin time (PT) and partial thromboplastin time (PTT) have to be within normal limits, unless the patient has been therapeutically anti-coagulated for previous venous thrombosis.

Exclusion Criteria:

* Female subjects of reproductive potential who are pregnant or lactating;
* Previous treatment with any gene therapy products or other form immunotherapy;
* Uncontrolled active infection.
* Active or latent chronic hepatitis B [detectable hepatitis B surface antigen (HBsAg)] or active hepatitis C (positive serology [hepatitis C virus Ab]) infection.
* HIV infection;
* History of allergy or hypersensitivity to study product excipients (human serum albumin, Dimethyl sulfoxide, and Dextran 40);
* Currently enrolled in other clinical trials;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-02 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events attributed to the administration of the chimeric antigen receptor T cells | 1 year
  Determine the toxicity profile of the chimeric antigen receptor T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Objective Response Rate | 1 year
  The objective response rate (ORR) is defined as the proportion of patients who achieve radiographic partial or complete response (PR or CR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guideline.
clinical activity of chimeric antigen receptor T cells | 28 days
  the number of infused chimeric antigen receptor T cells;

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, China

REFERENCES:
- [Derived] Lin Q, Ba T, Ho J, Chen D, Cheng Y, Wang L, Xu G, Xu L, Zhou Y, Wei Y, Li J, Ling F. First-in-Human Trial of EphA2-Redirected CAR T-Cells in Patients With Recurrent Glioblastoma: A Preliminary Report of Three Cases at the Starting Dose. Front Oncol. 2021 Jun 21;11:694941. doi: 10.3389/fonc.2021.694941. eCollection 2021. PMID 34235085